CLINICAL TRIAL: NCT02360657
Title: A Double-blind, Placebo-controlled, Randomized, 4-Week, Multiple-dose, Proof of Mechanism (POM) Study in Japanese Subjects Asymptomatic at Risk for Alzheimer Dementia (ARAD) Investigating the Effects of JNJ-54861911 on A-beta Processing in Cerebrospinal Fluid (CSF) and Plasma
Brief Title: Study Investigating the Effects of JNJ-54861911 on Amyloid-beta Processing in Cerebrospinal Fluid (CSF) and Plasma in Japanese Participants Asymptomatic at Risk for Alzheimer Dementia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR106397; 54861911ALZ1008 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2015-02-05; First posted 2015-02-10 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Alzheimer Dementia; JNJ-54861911; Beta Secretase Inhibitor
MeSH Terms: conditions — Alzheimer Disease | interventions — atabecestat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- JNJ-54861911, 10 mg (Experimental): JNJ-54861911, 10 milligram (mg) (2*5 mg tablet) orally once daily for 4 weeks.
  Interventions: Drug: JNJ-54861911, 10 mg
- JNJ-54861911, 50 mg (Experimental): JNJ-54861911, 50 mg (2*25 mg tablet) orally once daily for 4 weeks.
  Interventions: Drug: JNJ-54861911, 50 mg
- Placebo (Placebo Comparator): Placebo matching to JNJ-54861911 tablet orally once daily for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-54861911, 10 mg — JNJ-54861911, 10 mg (2*5 mg tablet) orally once daily for 4 weeks.
  Arms: JNJ-54861911, 10 mg
Drug: JNJ-54861911, 50 mg — JNJ-54861911, 50 mg (2*25 mg tablet) orally once daily for 4 weeks.
  Arms: JNJ-54861911, 50 mg
Drug: Placebo — Placebo matching to JNJ-54861911 tablet orally once daily for 4 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety, tolerability and effect of JNJ-54861911 on level of amyloid-beta in Cerebrospinal Fluid (CSF) and plasma following 4 weeks of treatment in Japanese participants asymptomatic at risk for Alzheimer Dementia (ARAD) at the intended target dose range.

DETAILED DESCRIPTION:
This is a multi-center (when more than one hospital or medical school team work on a medical research study), double-blind (neither physician nor participant knows the treatment that the participant receives), placebo-controlled (the experimental treatment or procedure is compared to an inactive substance), randomized (study medication assigned by chance), multiple dose, Proof of Mechanism (POM) study in Japanese participants ARAD. All eligible participants will be randomly assigned to 1 of 3 treatment groups (that is, placebo, JNJ-54861911 10 milligram [mg] or JNJ-54861911 50 mg once daily regimen). This study will consist of Screening Phase (8-week), Double blind Treatment Phase (4-week), and Follow-up Phase (2-week). The maximum study duration for a participant will be 14 weeks. Participant's safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have had sufficient education or work experience to exclude mental retardation based on Diagnostic and Statistical Manual of Mental Disorders 4th edition, Text Revision (DSM-IV-TR) and must be able to read and write and must have adequate hearing and visual acuity to complete the required psychometric tests
* Participant must have a Clinical Dementia Rating Scale- Japanese version (CDR-J) score of '0' and as such rated as normal
* Participant must have evidence of amyloid deposition as demonstrated by low Cerebrospinal Fluid (CSF) Amyloid (A)-beta 1-42 levels at Screening
* Participant must have a body mass index between 18 and 35 kilogram per square meter, inclusive, at Screening
* Participant must be otherwise healthy for their age group or medically stable with or without medication on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at Screening or at Baseline

Exclusion Criteria:

* Participant has evidence of any brain disease other than potential very early signs of Alzheimer's disease (AD) or typical age related changes, or any other abnormality that could explain a possible cognitive deficit
* Participant has been diagnosed with dementia due to AD, due to other diseases, or with AD and contribution of other disorders (mixed dementia)
* Participant has evidence of familial autosomal dominant AD
* Participant has any contra-indications for Magnetic Resonance Imaging (MRI) (for example, prostheses, implants, claustrophobia, pacemakers, and others)
* Participant has a clinically significant abnormal physical- or neurological examination, vital signs or 12-lead ECG (including QTc greater than 450 millisecond for males and females, left bundle branch block, atrio-ventricular [AV] block second degree or higher, permanent pacemaker or implantable cardioverter defibrillator [ICD]) at Screening or Baseline, which in the opinion of the investigator is not appropriate and reasonable for the population under study

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-02-16 (Actual); Primary Completion 2015-09-08 (Actual); Study Completion 2015-09-08 (Actual)

PRIMARY OUTCOMES:
Levels of Amyloid (A)-beta1-40 in Cerebrospinal Fluid (CSF) After Treatment at the Intended Target Dose Range | Up to 4 weeks
Levels of A-beta1-40 in Plasma After Treatment at the Intended Target Dose Range | Up to 4 weeks
Maximum Observed Plasma Concentration (Cmax) of JNJ 54861911 | Up to 4 weeks
  The Cmax is the maximum observed plasma concentration.
Minimum Observed Plasma Concentration (Cmin) of JNJ 54861911 | Up to 4 weeks
  The Cmin is the minimum observed plasma concentration.
Time to Reach Maximum Observed Concentration (Tmax) of JNJ 54861911 | Up to 4 weeks
  The Tmax is time to reach the maximum observed plasma concentration.
Area Under the Curve From Time Zero to end of Dosing Interval (AUCtau) | Up to 4 weeks
  The AUCtau is a measure of the plasma drug concentration from time zero to end of dosing interval. It is used to characterize drug absorption.
Cerebrospinal Fluid Exposure of JNJ-54861911 | Up to 4 weeks
The Number of Participants who Experienced Adverse Events as a Measure of Safety and Tolerability of JNJ-54861911 After Multiple-Dose Administration in the Anticipated Target Dose Range | Up to 4 weeks
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

SECONDARY OUTCOMES:
Levels of A-beta Fragments (A-beta1-37, A-beta1-38, and A-beta1-42) in CSF After Treatment at the Intended Target Dose Range | Up to 4 weeks
Levels of A-beta Fragments (A-beta1-37, A-beta1-38, and A-beta1-42) in Plasma After Treatment at the Intended Target Dose Range | Up to 4 weeks
Levels of Soluble Amyloid Precursor Protein (APP) Fragments in CSF (sAPP-alpha, sAPP-beta, totalAPP) After Treatment at the Intended Target Dose Range | Up to 4 weeks
Compare the Relationship of A-beta1-40 Levels in Plasma and CSF After Treatment at the Intended Dose Range | Up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (2):
- Japan (2):
  - Fukuoka
  - Tokyo

REFERENCES:
- [Derived] Timmers M, Streffer JR, Russu A, Tominaga Y, Shimizu H, Shiraishi A, Tatikola K, Smekens P, Borjesson-Hanson A, Andreasen N, Matias-Guiu J, Baquero M, Boada M, Tesseur I, Tritsmans L, Van Nueten L, Engelborghs S. Pharmacodynamics of atabecestat (JNJ-54861911), an oral BACE1 inhibitor in patients with early Alzheimer's disease: randomized, double-blind, placebo-controlled study. Alzheimers Res Ther. 2018 Aug 23;10(1):85. doi: 10.1186/s13195-018-0415-6. PMID 30134967